CLINICAL TRIAL: NCT00869687
Title: A Single Group Study for the Characterization of Human Tissue Response to Injectable Poly-L-Lactic Acid (Sculptra) in Healthy Volunteers
Brief Title: Biopsy Study for Sculptra (Poly-L-Lactic Acid)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: POLYL_L_02888
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Poly-L-Lactic Acid Injection (Other)
  Interventions: Device: Poly-L-Lactic Acid Injection

INTERVENTIONS:
Device: Poly-L-Lactic Acid Injection — 0.05 mL of poly-l-lactic acid will be injected as depot at three (3) points (a total of 0.15 mL).

SUMMARY:
The primary objective of this study involves research to evaluate new collagen (the elastic fibers that provide skin with its strength and resilience) formation in the skin following injections of Sculptra (Poly-L-Lactic Acid or PLLA). The secondary objectives of the study are to better understand the human skin responses to Sculptra and to assess the safety of Sculptra injections.

ELIGIBILITY:
Inclusion Criteria:

* If female, the subject must use appropriate form of birth control.

Exclusion Criteria:

* History of allergies or an allergic reaction to local numbing medications (e.g., lidocaine, etc.), latex, or silicone.
* History of forming large scars following an accident or surgery.
* History of any bleeding problems.
* Redness, swelling, or signs of infection behind the right or left ear between the area of the earlobe and hairline.
* Pimples, rashes, scarring or any other skin changes behind the right or left ear between the area of the earlobe and hairline.
* History of any medical problems (for example, heart attack, stroke, diabetes/high blood sugar, hepatitis, human immunodeficiency virus (HIV), severe asthma, rheumatoid arthritis, emphysema, breathing problems). Subjects with high blood pressure or high cholesterol may qualify for the study if there have been no changes in their medications for three (3) months.
* History of cancer within five (5) years.
* Previous cosmetic surgery or cosmetic procedures affecting the area behind the ear.
* Subject who plans to have any facial or ear surgery within the next year.
* History of alcohol or drug abuse.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Biopsies change from baseline to 6 months after first Sculptra injection in level of Type 1 collagen. | 6 months

SECONDARY OUTCOMES:
Change from baseline in level of Type 1 collagen at 3 months and 12 months | 3 and 12 months
Change from baseline in level of Type III collagen at 3 months, 6 months, & 12 months by immunohistochemistry in a central laboratory. | 3, 6, and 12 months
Qualitative assessment in degree of change from baseline in Type I collagen at 3 months, 6 months, & 12 months by a pathologist. | 3, 6, and 12 months
Degree of inflammation assessed by histology at 3 months, 6 months, and 12 months. | 3, 6, and 12 months
Qualitative assessment in degree of change from baseline in Type III collagen at 3 months, 6 months, & 12 months by a pathologist. | 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tara Semanchik, MBA, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Laval, Canada